CLINICAL TRIAL: NCT05499377
Title: Effects of Heated Tobacco Product Flavor on Tobacco Use Behavior and Abuse Liability Among Menthol Cigarette Smokers
Brief Title: The Abuse Liability of a Novel Heated Tobacco Product (IQOS) and Its Feasibility as a Menthol Cigarette Substitute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20024873; 1F30DA057047 (NIH); U54DA036105 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
Keywords: Heated Tobacco Products; Flavor; Abuse Liability; Tobacco; Cigarettes; Menthol; Experimental Tobacco Marketplace; Nicotine Delivery; Puff Topography; Ecological Momentary Assessment; Modified Risk Tobacco Product; IQOS; Heated Tobacco Products Flavors
MeSH Terms: conditions — Tobacco Use | interventions — Physical Examination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Tobacco-Flavored IQOS (Active Comparator): Tobacco - where menthol smokers will only have access to tobacco-flavored HeatSticks to use in the IQOS 2.4 Tobacco Heating System
  Interventions: Device: Tobacco product administration and assessment
- Menthol-Flavored IQOS (Experimental): Menthol - where menthol smokers will only have access to menthol-flavored HeatSticks to use in the IQOS 2.4 Tobacco Heating System
  Interventions: Device: Tobacco product administration and assessment

INTERVENTIONS:
Device: Tobacco product administration and assessment — Participants are first instructed to smoke their usual brand of menthol cigarettes normally for the next 7 days and avoid using any other tobacco products. After this baseline week, participants are randomized to 1 of 2 HTP flavor conditions (tobacco-flavored HeatSticks or Fresh Menthol-flavored HeatSticks), with equal probability and provided with a supply of their condition specific HTP and asked to use it in place of their usual menthol cigarettes for the next week. Participants use their own brand menthol cigarettes and assigned HTP both at home (naturalistic use) and in the clinical laboratory (two visits/week).

SUMMARY:
This project examines the influence of flavor availability on switching to an MRTP known as IQOS, part of the Heated Tobacco Product (HTP) class, among menthol smokers using clinical lab and naturalistic evaluations of abuse liability. Results will help federal regulators predict the public health impact on menthol cigarette smokers of policies restricting access to menthol-flavored HTPs.

DETAILED DESCRIPTION:
The public health success of FDA's proposed ban on menthol cigarettes hinges upon whether menthol smokers who are unable to quit smoking switch to non-menthol cigarettes (no public health gain) or to potentially lower harm alternatives like heated tobacco products (HTP). In 2019, FDA authorized an HTP called "IQOS" and its tobacco- and menthol-flavored "HeatSticks" (HS) as a modified risk tobacco product (MRTP). One issue relevant to FDA's future action regarding IQOS will be "whether and how certain flavors may help adult cigarette smokers reduce cigarette use and switch to potentially less harmful products" (FDA, 2018). Understanding the potential for HTPs like IQOS to reduce the health burden of cigarettes requires targeted research investigating the extent to which flavor availability is important for menthol smokers to switch to HTPs. For one tobacco product to substitute for another, their abuse liabilities should be congruent. Validated clinical lab methods exist for comparing tobacco product abuse liability by characterizing their nicotine delivery profiles (via plasma nicotine and puff topography) and reinforcing efficacy (via subjective and behavioral measures). Naturalistic assessment can validate clinical lab results regarding use patterns and product substitution.

The current study involves a two-arm, two-week, parallel group trial. The first week is an own brand (OB) menthol cigarette baseline, during which tobacco use will be assessed daily using ecological momentary assessment (EMA). On Monday and Friday, participants will complete clinical lab sessions that involve using OB cigarettes and responding to subjective measures and an Experimental Tobacco Marketplace (ETM) task that assesses willingness to substitute menthol cigarettes with an array of tobacco products including IQOS. During the next week, participants will be randomized to receive IQOS-menthol (n=25) or IQOS-tobacco (n=25); EMA and clinical lab visits will be repeated. Aim 1 assesses IQOS' abuse liability in a clinical lab setting. Outcomes include plasma nicotine levels, puffing behavior, responses about subjective effects, and product substitution from the ETM task. Aim 2 measures tobacco use patterns in naturalistic settings where participants will report daily OB and IQOS use outcomes via EMA. The overarching hypothesis is that, relative to OB, IQOS-menthol's abuse liability profile will differ less than IQOS-tobacco's, suggesting that menthol smokers will be more likely to substitute an HTP for combustible menthol cigarettes when a menthol-flavored HTP is available. Results will deepen our understanding of the public health impact of HTPs and policies that might restrict access to menthol-flavored MRTPs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (aged 21 and older)
* Daily menthol cigarette smokers
* Exhaled Carbon Monoxide (CO) reading of > 5 PPM at in-person screening (to confirm smoking status)
* A 'positive' cotinine cassette result to verify nicotine use at the in-person screening.
* Participants must be willing to provide informed consent and abstain from nicotine/tobacco for ≥8 hours prior to each lab session.
* Participants must have access to a computer/smartphone and be willing to receive and respond to daily surveys
* Able to read and write in English

Exclusion Criteria:

* Daily use of any tobacco products other than cigarettes
* Self-reported history of chronic medical or psychiatric conditions
* Women will be excluded if they test positive for pregnancy (by urinalysis) or self-report breastfeeding.

Some details of the study inclusion and exclusion criteria are omitted at this time, to preserve scientific integrity. Full inclusion and exclusion criteria will be posted following study completion.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Barnes, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White AM, Imran R, Gaitan N, Bickel WK, Perera RA, Cobb CO, Eissenberg TE, Barnes AJ. A Pilot RCT Exploring Heated Tobacco Product Substitution for Menthol Cigarettes. Am J Prev Med. 2025 Nov;69(5):108029. doi: 10.1016/j.amepre.2025.108029. Epub 2025 Aug 5. PMID 40763831

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Started | 15 | 18
Completed | 12 | 18
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 18 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.6) | 43.0 (8.3) | 44.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 13 | 22
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Average Daily Cigarette Use Per Day From Baseline
Description: Average number of cigarettes consumed per day, collected via daily text/email survey, averaged overconsumption for Tues-Thurs of each week. Outcome will compare the percent change in cigarette consumption from the baseline week (OB menthol cigarette use) to the intervention week (IQOS use) between the two study arms.
Time Frame: Week 1 (baseline) to Week 2 (intervention)
Population: Percent change in Average Daily Cigarette Use per day from baseline
Measure: Median (Inter-Quartile Range); unit: % reduction in cigarettes per day
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
% reduction in cigarettes per day | 36.8 [30.0 to 44.0] | 80.36 [46.7 to 89.2]

2. Primary Outcome: Percent Increase in Demand as the Subject is Willing to Substitute From Cigarettes to HTPs Using the Experimental Tobacco Marketplace Task
Description: Participants will complete the Experimental Tobacco Marketplace Task - which asks participants to allocate a hypothetical budget across a large menu of products. In each session, cigarette prices increased ($0.12, $0.25, $0.50, $1.00. and $2.00 per cigarette) while prices for alternative products remained fixed. Across three ETM sessions, either all products, all products except little cigars and cigarillos (LCCs), or all products except ENDS (JUUL e-cigarettes) were available. Linear regression is performed on individual participant data using log-transformed cigarette price to determine demand and substitution. Reported demand for tobacco products is used to determine substitution between IQOS and cigarettes. Purchasing decisions are not reinforced. Outcome will compare the cross-price elasticity (CPE) of IQOS with respect to menthol cigarettes among those with access to IQOS-menthol and IQOS-Tobacco (IQOS-M group) compared to those with access to IQOS-tobacco only (IQOS-T group).
Time Frame: Week 2, Friday Clinical Lab visit
Measure: Mean (Standard Deviation); unit: percent increase in demand/dollars
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
percent increase in demand/dollars | 0.14 (0.4) | 0.67 (0.8)

3. Primary Outcome: Plasma Nicotine Delivery
Description: Change in the plasma nicotine levels from before to after a standardized 10-puff (30-sec interpuff interval) bout with IQOS in the participant's assigned flavor. Outcome will compare the average plasma nicotine boost (the change in plasma nicotine levels from before to after the standardized puffing bout) across two study arms as well as compared to own-brand menthol cigarettes.
Time Frame: Week 2, Friday Clinical Lab visit (10 puff bout period)
Measure: Median (Inter-Quartile Range); unit: Nicotine boost (ng/mL)
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
Nicotine boost (ng/mL) | 6.3 [1.12 to 8.3] | 6.6 [0.4 to 7.7]

4. Secondary Outcome: Cigarette Craving Suppression Questionnaire
Description: We will compare the degree of "cigarette craving" will be assessed before and after a 10-puff use bout of IQOS. Cigarette craving will be assessed before and after a standardized puffing bout using the Questionnaire of Smoking Urges (QSU), which features 7-point likert-like scales. The reduction in "urges to smoke" item from the QSU will be used in this assessment. The average cigarette craving suppression score will be compared across the two experimental IQOS groups. The Tobacco Craving Questionnaire (TCQ) is a valid and reliable 47-item self-report instrument that assesses tobacco craving in four dimensions: emotionality, expectancy, compulsivity, and purposefulness. The higher your score, the more likely you are to have withdrawal symptoms if you give up smoking; also, the withdrawal symptoms are likely to be stronger
Time Frame: Week 2, Friday Clinical Lab Visit (10 puff bout period)
Measure: Median (Inter-Quartile Range); unit: change in craving (0-100) scale
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
change in craving (0-100) scale | -9.5 [-45.5 to 2] | -41.5 [-62 to -16]

5. Secondary Outcome: Puff Topography (Puff Duration)
Description: Average duration per puff during a standardized 10-puff (30-sec interpuff interval) bout with IQOS in assigned flavor. Puff duration will be measured using a validated puff topography instrument that attaches to the IQOS device. Outcome will compare the average puff duration across two study arms.
Time Frame: Week 2, Friday Clinical Lab visit (10 puff bout period)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
seconds | 1.64 [1.2 to 2.9] | 1.33 [1.1 to 2.1]

6. Secondary Outcome: Average Daily IQOS Usage
Description: Number of IQOS HeatSticks used each day will be assessed during the study. We will compare the number of Heatsticks used per day, on average (from Tues-Thurs of intervention week), between the two study arms.
Time Frame: Week 2 (intervention week), Tuesday-Thursday
Measure: Mean (Inter-Quartile Range); unit: IQOS sticks per day
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
Number analyzed (Participants) | 12 | 18
IQOS sticks per day | 4.5 [1.7 to 6.7] | 4.3 [3.3 to 9.7]

ADVERSE EVENTS:
Time Frame: Collected over the duration of participation (2 weeks) while study was active (10 months).
Arm/Group | Tobacco-Flavored IQOS | Menthol-Flavored IQOS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/12 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT05499377/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT05499377/ICF_001.pdf